CLINICAL TRIAL: NCT05182931
Title: A Prospective, Multi-Centre Trial of TKI Redifferentiation Therapy in Patients With RAIR Thyroid Cancer (I-FIRST Study)
Acronym: I-FIRST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Royal North Shore Hospital (Other); Austin Health (Other Government); Sir Charles Gairdner Hospital (Other); Monash Health (Other); Peter MacCallum Cancer Centre, Australia (Other); Royal Brisbane and Women's Hospital (Other Government); Eastern Health (Other); The Alfred (Other); Royal Adelaide Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2021-006
Record Dates: First submitted 2021-11-23; First posted 2022-01-10 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Cancer
Keywords: Radioiodine refractory; BRAF600E mutant; RAS mutant
MeSH Terms: conditions — Thyroid Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Participants with BRAF V600E mutant thyroid cancer will receive Dabrafenib + Trametinib; Participants with RAS mutant thyroid cancer will receive Trametinib alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BRAFv600E mutant radioiodine refractory thyroid cancer (Experimental): Prior to commencing interventional treatment, participants will commence a low iodine diet and undergo thyroxine withdrawal and commence T3 replacement from day -27. On day -5 they will receive an oral dose of 124I (40MBq/1.08 mCi) with imaging at 24 hours (+/-6) post dose and a second imaging assessment within 120 hours.
  Participants will receive Dabrafenib (oral, 150mg BD) and Trametinib (oral, 2mg OD) from day 1-30.
  A second oral dose of I124 will be administered at day 24 followed by imaging at the same interval as baseline.
  Participants achieving >20Gy tumour uptake of I124 will be administered 6GBq (3.3Gy/GBq) 131I, I131 wb scan and SPECT/CT will be performed within 24 hours and at hospital discharge.
  Participants who do not achieve >20Gy tumour update of I-124 will move into follow up.
  Follow up will occur every 12 weeks for 12 months.
  Interventions: Drug: Dabrafenib 75 MG; Drug: Trametinib 2 MG
- RAS mutant radioiodine refractory thyroid cancer (Experimental): Prior to commencing interventional treatment, participants will commence a low iodine diet and undergo thyroxine withdrawal and commence T3 replacement from day -27. On day -5 they will receive an oral dose of 124I (40MBq/1.08 mCi) with imaging at 24 hours (+/-6) post dose and a second imaging assessment within 120 hours.
  Participants will receive Trametinib (oral, 2mg OD) from day 1-30.
  A second oral dose of I124 will be administered at day 24 followed by imaging at the same interval as baseline.
  Participants achieving >20Gy tumour uptake of I124 will be administered 6GBq (3.3Gy/GBq) 131I, I131 wb scan and SPECT/CT will be performed within 24 hours and at hospital discharge.
  Participants who do not achieve >20Gy tumour update of I-124 will move into follow up.
  Follow up will occur every 12 weeks for 12 months.
  Interventions: Drug: Trametinib 2 MG

INTERVENTIONS:
Drug: Dabrafenib 75 MG — Refer arm description
  Other Names: Tafinlar
  Arms: BRAFv600E mutant radioiodine refractory thyroid cancer
Drug: Trametinib 2 MG — Refer arm description
  Other Names: Mekinist

SUMMARY:
This prospective, multi-centre, open label, non-randomised phase II trial aims restore radioiodine sensitivity in patients with NRAS or BRAFV600E mutant refractory thyroid cancer.

Participants will be treated with Trametinib +/- Dabrafenib tyrosine kinase inhibitors for a period of 30 days, restoration of sensitivity will be monitored using 18F-FDG-PET & I-124 PET imaging.

DETAILED DESCRIPTION:
This is a prospective, non-randomised, multi-centre study which will be conducted at 10 sites around Australia.

Adult patients (18+ years) with radioiodine refractory differentiated thyroid cancer with BRAF V600E or NRAS mutant RECIST 1.1 evaluable tumours will be eligible to participate. .

All eligible patients will undergo a 18F-FDG PET/CT scan during the registration period (day -28), followed by T4 withdrawal and low iodine diet. T3 will be administered after T4 withdrawal and for up to 10 days prior to the 124I dose to minimise symptoms of hypothyroidism.

The first 124I dose will be administered orally at a dose of 40 MBq (1.08 mCi) on day -5 with a 18FDG-PET performed on the same day. Patients will then have 124I-PET imaging and bloods at 24 hrs (+/- 6 hrs) post-dose, with a second imaging time-point up until 120 hours post- 124I dose. The initial 124I study (pre-TKI) will serve as a baseline for the second 124I-PET (day 24, after 23 days of TKI), and demonstrate changes in NIS expression and radioiodine uptake as a result of TKI treatment.

Patients will then commence a total of 30 days of treatment with the MEK TKI trametinib (for NRAS mutant tumours) or the MEK and BRAF V600E TKI combination of trametinib and dabrafenib (for BRAF V600E mutant tumours). Patients will then have a further 18F-FDG PET/CT scan and 124I dose on day 23, and scans for dosimetry (124I-PET) at 24 hrs (+/- 6 hrs) post-dose (day 24), with a second imaging time-point up until 120 hours post-124I administration. If at least one lesion shows uptake on 124I scans consistent with > 20Gy / 6GBq (3.3Gy/GBq) 131I administered (based on the 24-hour scan), then 131I treatment will be administered on day 29. The dose of 131I administered will be fixed at 6 GBq (150 mCi) to allow for evaluation of dose response. TKI treatment will continue until the day after 131I treatment is given (total 30 days).

Follow-up staging (CT) will occur every 3 months for the first 24 months, then every 6 months until progression, and 18F-FDG PET at 6 and 12 months. Non-stimulated thyroglobulin (Tg) will also be measured at 3, 6, 9 and 12 months, and evaluated as a percentage change from baseline. QoL and health economic data will be collected in all patients going on study. Overall survival will be obtained by long-term follow-up. Central review of tumour mutations, 124I PET dosimetry, staging (RECIST) and 18F-FDG PET (PERCIST) will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed differentiated (including poorly differentiated) thyroid cancer that is either locally advanced or metastatic.
2. Age > 18 years.
3. Life expectancy > 12 weeks.
4. Documented radiological progression by RECIST 1.1 in last 12 months.
5. Radioiodine refractory (at least one of):

   1. one measurable lesion without radioiodine uptake on 131I scan,
   2. at least one measurable lesion that had progressed by RECIST criteria within 12 months of 131I therapy despite 131I avidity at time of treatment, or
   3. cumulative treatment with >24 GBq (600 mCi) of 131I.
6. At least one evaluable lesion as per RECIST v1.1 that has not been treated with local radiation therapy within 3 months prior to the first dose of TKI. Irradiated lesions can only be included as an evaluable lesion if it has shown radiological progression as per RECIST v1.1 on subsequent imaging following irradiation.
7. NRAS or BRAF V600E mutation tested by NGS in a NATA accredited laboratory or by recognised sequencing platform.
8. ECOG 0-1.
9. Informed consent.
10. Adequate haematological and biochemical parameters:

    1. Haemoglobin ≥ 9g/dL
    2. Neutrophils ≥ 1.5 x 109/L
    3. Platelets ≥ 100 x 109/L
    4. INR ≤ 1.4
    5. Serum Creatinine ≤ 1.3 x ULN
    6. Estimated Creatinine Clearance ≥ 30 ml/min (by Cockcroft Gault Formula)
    7. Serum ALT and AST ≤ 2.5 x ULN
    8. Serum Total Bilirubin ≤ 1.5 x ULN.
    9. TSH suppression <0.1mU/L or otherwise consistent with 2015 ATA Guidelines on Thyroid Cancer

Exclusion Criteria:

1. Anaplastic thyroid cancer.
2. Suitable for curative surgery or radiotherapy.
3. Other anti-cancer (including TKI) therapy in prior 6 weeks.
4. Concurrent malignancy other than non-melanoma skin cancer. Prior malignancies treated with curative intent and no evidence of recurrence in past three years may be allowed upon discussion with the medical monitor.
5. Unstable brain metastasis. Treated or non-treated brain metastasis are allowed if neurologically stable, asymptomatic, on a stable steroid dose for a period of 2 weeks, and not anticipated to require any intervention during the trial treatment period. If treated with radiation or surgery, any related AE's should have recovered to ≤ grade 1 prior to enrolment on trial.
6. Pregnancy, breastfeeding or unwilling to use contraception in those of child-bearing age.
7. Significant medical condition that would prevent compliance with study procedures.
8. History of retinal vein occlusion or retinopathy.
9. Iodine-containing contrast scan within 8 weeks of planned 124I scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival as assessed by RECIST 1.1 criteria at 6 months in participants who proceed to I131 treatment | At 6 months following day 1.
  Radioiodine refractory thyroid cancer patients able to proceed to 131I treatment will be assessed by RECIST 1.1 criteria.
Progression free survival as assessed by RECIST 1.1 criteria at 12 months in participants who proceed to I131 treatment | At 12 months following day 1.
  Radioiodine refractory thyroid cancer patients able to proceed to 131I treatment will be assessed by RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression free survival as assessed by RECIST 1.1 criteria at 6 months in all participants and a control population (SELECT study) | At 6 months following day 1.
  To assess PFS by RECIST v1.1 at 6 in radioiodine-refractory thyroid cancer patients able to proceed to 131I treatment following TKI redifferentiation therapy,
  1. compared to those who do not proceed to 131I treatment.
  2. compared to a control population (from the SELECT study).
Progression free survival as assessed by RECIST 1.1 criteria at 12 months in all participants and a control population (SELECT study) | At 12 months following day 1.
  To assess PFS by RECIST v1.1 at 12 months in radioiodine-refractory thyroid cancer patients able to proceed to 131I treatment following TKI redifferentiation therapy,
  1. compared to those who do not proceed to 131I treatment.
  2. compared to a control population (from the SELECT study).
Objective response rate by RECIST 1.1 criteria in all treated participants | 0-18 months or at PD
  To assess objective response (CR/PR/SD) in all treated participants from time of enrolment until 18 months or PD.
Overall survival of treated participants | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  To confirm the overall survival of participants receiving treatment on study via Kaplan-Meier estimation.
Quantification of treatment related toxicities according to CTCAE V5.0 | From day -27 until 30 days following last dose [up to max 60 days].
  Quantification of treatment related toxicities according to CTCAE V5.0
Quantification of radioiodine uptake in metastatic lesions before and after TKI treatment. | From day -5 until day 30 on study.
  Quantification of radioiodine uptake in metastatic lesions before and after TKI treatment.
Evaluation of response to treatment by percent change from baseline of non-stimulated thyroglobulin. | Day 0; 3, 6, 9, 12 months in participants without radiological progression.
  Evaluation of response to treatment by percent change from baseline of non-stimulated thyroglobulin.
Evaluation and comparison of quality of life as measured by response to EORTC-QLQ-C30 in participants on study. | Day -29, 1, 29; 3, 6, 9, 12 months.
  Evaluation of QOL in participants who proceed to I131 treatment compared with participants who proceed to follow up only by EORTC-QLQ-C30. Scores are from 0-100 with participant reported quality of live improving with a higher score.
Evaluation and comparison of QOL as measured by response to EQ-5D-5L in participants on study. | Day -29, 1, 29; 3, 6, 9, 12 months.
  In participants who proceed to I131 treatment compared with follow up only by EQ-5D-5L. Five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems to extreme problems.
Evaluation and comparison of QOL as measured by response to Kessler Psychological Distress Scale (K10) in participants on study. | Day -29, 1, 29; 3, 6, 9, 12 months.
  In participants who proceed to I131 treatment compared with follow up only by responses to the Kessler Psychological Distress Scale (K10). This is a 10-item questionnaire yielding a global measure of distress based on questions about anxiety and depressive symptoms. 5 levels ranging from none of the time to all of the time, higher level responses correspond with greater reported distress.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Scott, MD, FRACP, Study Chair — Austin Health
Locations (9):
- Australia (9):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hsopital, Adelaide, South Australia
  - Eastern Health, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Peter MacCallum Cancer Centre, Melbourne

IPD SHARING:
Plan to Share IPD: No